CLINICAL TRIAL: NCT06332989
Title: Comparison of Prehospital Stroke Screening Scales in the Ambulance Setting; a Multiregional, Multicenter Observational Cohort Study
Brief Title: Stroke Triage Optimization by Ambulance Paramedics in the Pre-hospital Setting
Acronym: STROKE-APP
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Alrijne Ziekenhuis Leiderdorp (Network); Groene Hart Ziekenhuis (Other); Medical Center Haaglanden (Other); HagaZiekenhuis (Other); Reinier de Graaf Groep (Other); Regionale Ambulance Voorziening Hollands Midden (Other)
Responsible Party: Principal Investigator, NyikaKruyt, M, PhD, Leiden University Medical Center
Other Study IDs: N22.129
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Stroke, Acute; Pre-hospital Triage; Stroke Treatment; Stroke Code
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: stroke-APP — Ambulane paramedics will use an online application to fill in several observations on scen

SUMMARY:
There are everal scales designed to help ambulance paramedics to identify a patient with a stroke and activate a stroke code. These scales were never tested in the field in a large unselected patient sample. We aim to perform an in-the field head tot head comparison of all published stroke scales designed to be used by ambulance paramedics

DETAILED DESCRIPTION:
this is a multicenter multiregional cohort study including about 3000 stroke code patients. In all patients an application will be filled out before hospital arrival including items that enable us to reconstruct all previously published stroke scales.

Data from the application will be related to in hospital data of the same patient. In order to do this we will use a trusted third party for data coupling.

ELIGIBILITY:
Inclusion Criteria:

* patients for whom a stroke code is activated

Exclusion Criteria:

< 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients for whom a stroke code was activated.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
final diagnosis | discharge or after 3 months
  Diangosis by treating physician
treated with reperfusion therapy | first 24 hours after admission
  treatment with IV thrombolysis; endovascular therapy or surgery
additional investigations | on admission
  CT scans performed

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University medical center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided